CLINICAL TRIAL: NCT01163669
Title: A Prospective Cohort Study to Describe the Evolution of Persistent Hyperparathyroidism in Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20080093
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2012-01

CONDITIONS: Hyperparathyroidism
Keywords: hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- kidney transplant recipients

SUMMARY:
The purpose of this study is to see if Hyperparathyroidism (HPT) is common in people who receive a kidney transplant. Patients with HPT often have high parathyroid hormone (PTH) levels and may have large parathyroid glands in the neck. Patients with HPT can develop bone disease (osteodystrophy). This bone disease can cause bone pain, fractures, and poor formation of red blood cells. Other problems from HPT may include increases in blood levels of calcium (hypercalcemia) and low blood levels of phosphorus (hypophosphatemia). The high calcium levels may cause calcium to deposit in body tissues. Calcium deposits can cause arthritis (joint pain and swelling), muscle inflammation, itching, gangrene (death of soft tissue), heart and lung problems, or kidney transplant dysfunction (worsening of kidney transplant function). The purpose of this research study is to better understand the evolution of Hpt in people during the first 12 months after receiving a kidney transplant.

DETAILED DESCRIPTION:
Subjects are enrolled in the study and a 12-month observational phase will begin. During the observational phase, subjects will attend a total of 8 visits at approximately 1, 2, 4, and 8 weeks after kidney transplantation and at 3, 6, 9, and 12 months after kidney transplantation. During these visits, subjects will have a review of medication history, blood tests, and a kidney function test. The blood will be used to test the level of certain components of you blood to see if your HPT has resolved, stabilized, or advanced. At selected visits throughout the study, you will have a urine sample collected and a health questionnaire that will ask about your health. Information regarding transplant kidney biopsy (if performed) also will be collected.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CKD receiving hemodialysis prior to transplant;
* admission for kidney transplant surgery;
* men and women at least 18 year of age;
* one or more plasma PTH values determined during during the 6 months before screening that is greater the 65pg/ml;
* plasma PTH greater than 65pg/ml at screening before kidney transp[lant as measured by the central lab.

Exclusion Criteria:

* history of medical conditions that cause hypercalcemia such as primary HPT, active malignancy, and granulomatous diseases.
* receipt of multiple organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
plasma parathyroid hormone(PTH)level | 12 months

SECONDARY OUTCOMES:
corrected total serum calcium and phosphorus concentration | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: T Srinivas, MD, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States